CLINICAL TRIAL: NCT01276366
Title: Amphia Premature Infant Pain Study; Breast Milk vs Sucrose
Brief Title: Amphia Premature Infant Pain Study
Acronym: APIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amphia Hospital (Other)
Responsible Party: Principal Investigator, R.H.T. van Beek, dr. R.H.T. van Beek, Amphia Hospital, pediatric department, Amphia Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL30111.101.09
Record Dates: First submitted 2010-04-23; First posted 2011-01-13 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Premature Infant; Breast Feeding, Exclusive; Puncture Skin
Keywords: Heel lance; Premature; Breast milk
MeSH Terms: conditions — Premature Birth; Breast Feeding | interventions — Lactation; Sucrose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- sucrose (Active Comparator): In the third group, newborns receive sucrose 1ml 24% two minutes before procedure, followed by non-nutritive sucking. During the procedure the newborn lies in his cot.
  Interventions: Other: sucrose
- supplemental breast milk (Active Comparator): In group two, the newborns receive supplemental breast milk, lying in the arms of a nurse during the heel lance.
  Interventions: Other: supplemental breast milk
- Breast feeding (Active Comparator): Newborns who are assigned to group one, receive breastfeeding during the blood sample and thereby have skin-skin contact between mother and child.
  Interventions: Other: breast feeding

INTERVENTIONS:
Other: breast feeding — Newborns who are assigned to group one, receive breastfeeding during the blood sample and thereby have skin-skin contact between mother and child.
  Arms: Breast feeding
Other: supplemental breast milk — In group two, the newborns receive supplemental breast milk, lying in the arms of a nurse during the heel lance.
  Arms: supplemental breast milk
Other: sucrose — In the third group, newborns receive sucrose 1ml 24% two minutes before procedure, followed by non-nutritive sucking. During the procedure the newborn lies in his cot.
  Arms: sucrose

SUMMARY:
Last thirty years, many research was performed concerning pain in the newborn. These investigations showed us the negative effects of pain in the neonatal period. Our research concerns the choice of analgesics for the premature newborn during a heel lance. Newborns with a gestational age of 32-37 weeks are randomly assigned over three groups. They can receive breastfeeding, during the heel lance, a bottle with supplemental breast milk or sucrose.

The primary objective of the Amphia Premature Infant Pain study, is to investigate whether there is a difference in PIPP-scores in premature newborns who undergo a heel lance, receiving breast milk or sucrose. Our hypothesis is that the PIPP-score will be lower in newborns receiving breast milk compared to sucrose. And the investigators presume that breast feeding has the same analgesic effect as giving supplemental breast milk.

ELIGIBILITY:
Inclusion Criteria:

* born at a gestational age between 32+0 and 36+6 weeks,
* being nourished with breast milk
* the necessity for a clinical blood sample.

Exclusion Criteria:

* perinatal asphyxia,
* birth trauma,
* condition of cardio-respiratory instability,
* condition of serious nutritional problems with clinical evidence of gastro oesophageal reflux disease,
* drug abuse of the mother
* and application of sedative medication to mother or child.

Ages: 1 Day to 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2010-01-01; Primary Completion 2011-08-01 (Actual); Study Completion 2012-04-01 (Actual)

PRIMARY OUTCOMES:
Pain scores assessed by the PIPP score | The PIPP score will be assessed during a heellance. This heellance will be performed after one day of life and before two months.
  The primary outcome in this trial is the PIPP-score.The PIPP-score is a multidimensional pain assessment measure developed in 1995 . The PIPP-score is validated for procedural and post-operative pain in premature and term newborns.

SECONDARY OUTCOMES:
Pain score assessed by the COMFORTneo score | The COMFORTneo score will be assessed during a heellance. This heellance will be performed after one day of life and before two months.
  The COMFORTneo is a secondary outcome.The COMFORTneo is a pain assessment measure modified from the COMFORT behaviour scale. In 2009 the COMFORTneo is validated for prolonged pain. The COMFORTneo is not validated for procedural pain yet .
partial correlation between the two pain assessment tools. | up to 2 years
  A secondary outcome is the partial correlation between the PIPP-score and the COMFORTneo score for a heellance in babies born with a postconceptional age between 32 and 37 weeks. When all films are observed, the COMFORTneo scores and PIPP scores are evaluated. We measure a partial correlation coefficient between these scores, to compare these two scores.
intra-class correlation coefficient | up to 2 years
  This secondary outcome measure gives us information about the uniformity of the assessment of the films between the three investigators.

CONTACTS AND LOCATIONS:
Overall Officials: RHT v Beek, phd, Principal Investigator — Amphia Hospital Breda
Locations (1):
- Amphia Hospital, Breda, North Brabant, Netherlands

REFERENCES:
- [Derived] Simonse E, Mulder PG, van Beek RH. Analgesic effect of breast milk versus sucrose for analgesia during heel lance in late preterm infants. Pediatrics. 2012 Apr;129(4):657-63. doi: 10.1542/peds.2011-2173. Epub 2012 Mar 5. PMID 22392168